CLINICAL TRIAL: NCT04704752
Title: Clinical Characteristics of Swallowing in Pediatric Patients With Eosinophilic Esophagitis
Brief Title: Swallowing Characteristics of Pediatric Patients With Eosinophilic Esophagitis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, PhD, Gazi University
Other Study IDs: 888819
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Swallowing Evaluation — Study Evaluation includes basic test batteries. These are observational.

SUMMARY:
Eosinophilic Esophagitis (EoE) can affect patients all age group and clinical symptoms of the disease varies depending on the patient's ages. Infants and toddlers with EoE generally have food refusal, vomiting and poor weight gain. Older school-aged children and adolescents may have abdominal and chest pain, difficulty in swallowing (dysphagia) especially in solid foods. In the meantime, many children especially infants and toddlers, are not perceptive of their dysphagia, because they have the ability to compensate. Such as, avoiding certain textures or increases liquid intake in the meal.To date, to our knowledge, there is no study in the literature has investigated complex swallowing behaviour (including all phases), oral-motor evaluation and/or swallowing safety. Thus, the present study purposed to investigate (a) descriptive and clinical swallowing characteristics of children with EoE (b) the relation between disease characteristic and swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 2-17 years with a diagnosis of Eosinophilic Esophagitis

Exclusion Criteria:

* Do not accommodate the study
* Do not want to attempt the study

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescents aged 2-17 years with a diagnosis of Eosinophilic Esophagitis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Mastication and Observation Evaluation | 15 minutes
  Each child was positioned in an upright sitting position in a quiet environment. A standardized biscuit was offered in front of their mouth to bite and chew. Chewing performance of each child was scored according to the T-MOE by observing the child.

SECONDARY OUTCOMES:
Pediatric version of the Eating Assessment Tool-10 | 10 minutes
  The PEDI-EAT-10 is a parent report outcome instrument to determine penetration and aspiration risk in children.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, PhD, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation Recruiting Ankara, Turkey, 06500, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided yet.